CLINICAL TRIAL: NCT05112445
Title: Retinal Ischemia Characterization in Diabetes.
Brief Title: Retinal Ischemia Characterization in Diabetes - "RICHARD"
Acronym: RICHARD
Status: Active, not recruiting | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 4C-2021-10
Record Dates: First submitted 2021-10-20; First posted 2021-11-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retinal ischemia characterization in diabetes - RICHARD

DETAILED DESCRIPTION:
RICHARD is a non-interventional observational cross-sectional and prospective study. Patients will attend their routine clinical appointments, with 2-years of follow-up. Type 2 diabetic individuals with retinopathy ETDRS DRSS grade 43 with IRMA or grade 47-53 will be recruited and examined using non-invasive methodologies.

The study will be performed at AIBILI Clinical Trials Centre (CEC). Demographic and systemic parameters, such as diabetes duration, medical history, medication, body mass index, and family history of medical conditions (particularly when related to cognitive decline) will be registered at baseline.

All subjects will undergo an annual complete non-invasive ophthalmological examination, which includes, best corrected visual acuity, 7-fields CFP to assess ETDRS DRSS level, structural SD-OCT, SD-OCTA, SS-OCTA and ultra-widefield fundus photography (UWF FP). An invasive ophthalmological examination, the Ultra-wide field fundus fluorescein angiography (UWF FFA) will be obtained from both eyes at baseline (V0, M0) only in subjects with ETDRS DRSS grade 43 for final eligibility (43+IRMA).

Ophthalmological examinations performed will be analyzed at AIBILI Coimbra Ophthalmology Reading Centre (CORC) and Centre for New Technologies e Medicine (CNTM).

Color fundus photography (7-fields) will be acquired at V0 (month 0, baseline, cross-sectional study), V2 (month 12) and V3 (month 24), and then graded and classified according to the ETDRS severity scale by CORC, to allow evaluation of retinopathy progression over two years of follow-up. . At baseline visit (V0) both eyes will be evaluated and the study eye will be selected according to ETDRS DRSS grade (43 with IRMA, 47 or 53). Only the study eye will be considered for the primary statistical analysis; other statistical analyses will include both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 according to 1985 WHO definition.
* Age over 18 years old.
* NPDR levels ETDRS DRSS (43 with IRMA, 47 or 53), based on the ETDRS criteria - 7 fields CFP and UWF FFA for 43 with IRMA after confirmation by the Reading Centre (CORC).
* Refraction with a spherical equivalent less than 5 diopters
* Able to provide informed consent.

Exclusion Criteria:

* Presence of diabetic macular edema (DME) involving the center of the macula in the study eye and needing immediate treatment.
* Presence of CI-DME defined as central subfield thickness on OCT ≥305 µm if male or ≥290 µm if female on Zeiss Cirrus OCT [12] with vision loss and needing immediate treatment.
* Cataract or other eye disease that may interfere with fundus examinations or OCT/OCTA signal strength.
* Age-related macular degeneration, glaucoma, vitreomacular disease, other retinal vascular disease, or any ocular condition that, in the opinion of the investigator may affect retinopathy status or alter VA during the study.
* Any eye surgery, including laser, and anti-VEGF within a period of 6-months.
* Dilatation of the pupil > 5 mm.
* HbA1c > 12% in the last measurement prior to the study visit (V0). Study Eye: Only one eye per subject will be considered for the primary statistical analysis (Study Eye). If both eyes meet the inclusion criteria the study eye will be the one that has a higher level of DR (ETDRS classification). If both eyes have the same ETDRS DRSS grading, the eye with higher BCVA will be chosen. If both eyes have the same BCVA, the right eye will be chosen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 individuals with type 2 diabetes and diabetic retinopathy with ETDRS DRSS grade 43 with IRMA, 47 or 53, with or without previous treatment, will be included in this study, over a recruitment period of 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
OCTA metrics and predict progression to PDR and/ or CI- DME | Change from baseline to Month 12
  Identify which baseline OCTA metrics and predict progression to PDR and/ or CI- DME best correlate with visual function.
OCTA metrics and predict progression to PDR and/ or CI- DME | Change from baseline to Month 24
  Identify which baseline OCTA metrics and predict progression to PDR and/ or CI- DME best correlate with visual function.

CONTACTS AND LOCATIONS:
Locations (1):
- AIBILI-CEC (AIBILI- Clinical Trials Centre), Coimbra, Portugal

REFERENCES:
- [Derived] Marques IP, Reste-Ferreira D, Santos T, Mendes L, Martinho AC, Yamaguchi TCN, Santos AR, Pearce E, Cunha-Vaz J. Progression of Capillary Hypoperfusion in Advanced Stages of Nonproliferative Diabetic Retinopathy: 6-month Analysis of RICHARD Study. Ophthalmol Sci. 2024 Oct 16;5(2):100632. doi: 10.1016/j.xops.2024.100632. eCollection 2025 Mar-Apr. PMID 39639890
- [Derived] Santos AR, Lopes M, Santos T, Reste-Ferreira D, Marques IP, Yamaguchi TCN, Miranda T, Mendes L, Martinho ACV, Pearce L, Cunha-Vaz J. Intraretinal Microvascular Abnormalities in Eyes with Advanced Stages of Nonproliferative Diabetic Retinopathy: Comparison Between UWF-FFA, CFP, and OCTA-The RICHARD Study. Ophthalmol Ther. 2024 Dec;13(12):3161-3173. doi: 10.1007/s40123-024-01054-2. Epub 2024 Oct 26. PMID 39460896